CLINICAL TRIAL: NCT03918551
Title: Single Dose Crossover Comparative Bioavailability Study of Febuxostat 120 mg Film-Coated Tablets in Healthy Adult Subjects / Fasting State
Brief Title: Bioequivalence Study of Two Formulations of Febuxostat 120 mg Film-coated Tablets in Healthy Adult Volunteers After a Single Oral Dose Administration Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PTL-P1-099 (v. 1.0 03/15/2019)
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Bioequivalence
Keywords: bioequivalence; febuxostat; Adenuric
MeSH Terms: interventions — Febuxostat

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The randomization code will not be available to the personnel of the bioanalytical facility until the bioanalytical tables have been finalized and audited by the Quality Assurance (QA) department.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Other): 25 subjects assigned to the sequence AB will receive a single 120 mg dose of the test product Febuxostat (1 x 120 mg film-coated tablet), marked as A in the sequence, in Period 1 and a single 120 mg dose of the reference product Adenuric (1 x 120 mg film-coated tablet), marked as B in the sequence, in period 2. These treatments will be administered orally with approximately 240 mL of water at ambient temperature, in the morning, following a minimum of 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Febuxostat; Drug: Adenuric
- Sequence BA (Other): 25 subjects assigned to the sequence BA will receive a single 120 mg dose of the reference product Adenuric (1 x 120 mg film-coated tablet), marked as B in the sequence, in Period 1 and a single 120 mg dose of the test product Febuxostat (1 x 120 mg film-coated tablet), marked as A in the sequence, in period 2. These treatments will be administered orally with approximately 240 mL of water at ambient temperature, in the morning, following a minimum of 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Febuxostat; Drug: Adenuric

INTERVENTIONS:
Drug: Febuxostat — Febuxostat is manufactured by Pharmtechnology LLC, Republic of Belarus. Each film-coated tablet contains 120 mg of febuxostat.
  Other Names: the test product
Drug: Adenuric — Adenuric is manufactured by Menarini - Von Heyden GmbH, Germany (MAH: Menarini International Operations Luxembourg S.A., Luxembourg). Each film-coated tablet contains 120 mg of febuxostat.
  Other Names: the reference product

SUMMARY:
This study is designed in accordance with the European Medicines Agency (EMA) regulatory guidelines, with the aim of characterizing the bioavailability of febuxostat in the two formulations in healthy adult subjects. Within the clinical portion of the study each subject will receive a single oral dose of the test and the reference formulation in compliance with the generated randomization code. The primary study endpoints are the pharmacokinetic (PK) parameters Cmax and AUC0-T of febuxostat.

DETAILED DESCRIPTION:
This is a single center, randomized, 2-treatment, 2-period, 2-sequence, crossover, single dose study design, in which 50 healthy adult subjects will receive one of the study treatments during each study period.

The objective of this study is to determine the bioequivalence of two different formulations of febuxostat after a single oral dose administration under fasting conditions.

The intra-subject variation following a single dose of febuxostat appears to be up to 34% for Cmax and up to 12% for AUC0-T. Statistically, given that the expected Test to Reference ratio of geometric LSmeans should fall within 95 and 105%, it is estimated that the lowest number of subjects to meet the 80 to 125% bioequivalence range with a statistical a priori power of at least 80% is about 46. Therefore, the inclusion of 50 subjects should be sufficient to account for the possibility of drop-outs, variations around the estimated intra-subject CV and to conclude in favor of the hypothesis of bioequivalence with sufficient statistical power.

Subject eligibility for this study will be determined at the screening visit and eligible subjects will be admitted to the clinical research unit at least 10 hours prior to drug administration for each study period.

A subject who withdraws or is withdrawn during the pretrial evaluations but before receiving the investigational product (IP) will not be considered as a drop-out and will not be included in the final database. Standbys should be recruited and available to replace any subject who withdraws prior to the first drug administration. On-study drop-outs will not be replaced.

Altasciences will generate the randomization code with a computer program according to the study design, the number of subjects and the sequence of treatment administration. The random allocation of each sequence of treatment administration to each subject will be done in such a way that the study is balanced. Once generated, the randomization code will be final and will not be modified. Eligible subjects will be randomized to one of two treatment sequences. There will be two sequences in the study: AB and BA, where A = the test product, B = the reference product (see detailed description of A and B items in Section "Arms and Interventions").

For each study period, subjects will receive a single 120 mg oral dose of febuxostat (the test or the reference formulation), with approximately 240 mL of water at ambient temperature, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken. Study participants will be aware they will receive different formulations of the same drug, without being informed which product (Test or Reference) is being administered. The date and time of each dose will be recorded. For each subject, all scheduled postdose activities and assessments will be performed relative to the time of study drug administration.

Fasting will continue for at least 4 hours following drug administration, after which a standardized lunch will be served. A supper and a light snack will be served at appropriate times thereafter, but not before 9 hours after dosing. Water will be provided as needed until 1 hour predose. Water will be allowed beginning 1 hour after the administration of the drug.

In each study period, 21 blood samples will be collected for PK assessments. The first blood sample will be collected prior to drug administration while the others will be collected up to 36 hours after drug administration. Febuxostat plasma concentrations will be measured by a validated bioanalytical method.

Subjects are to be discharged from the clinic after the 36-hour postdose PK sample collection, and following medical approval. However, they may be advised to stay at the clinical site for safety reasons, if judged necessary by the physician in charge.

The expected terminal elimination half-life observed after a single oral 120 mg dose of febuxostat film-coated tablets under fasting conditions is 5.1 hours. To avoid any carry-over effect, a wash-out of 7 calendar days is planned between drug administrations.

The decision of which subjects will be included in the PK analysis is to be documented by the pharmacokineticist (or delegate) and approved by the sponsor before the start of the sample analysis by the bioanalytical facility. Subjects who are expected to provide evaluable PK data for both the Test and Reference products (based on viable PK samples) will be included in the pharmacokinetic analysis. Concentration data of the remaining subjects will be presented separately. Subjects who do not complete the sampling schedule of one or more study periods may be included in the PK and statistical analysis and bioequivalence determination for only the PK parameters that are judged not to be affected by the missing sample(s).

Statistical analysis of Tmax will be based on a non-parametric approach. Statistical analysis of all other pharmacokinetic parameters will be based on an analysis of variance (ANOVA) model. Two-sided 90% confidence interval of the ratio of geometric least-squares means (LSmeans) obtained from the ln-transformed pharmacokinetic parameters will be calculated.

Statistical inference of febuxostat will be based on a bioequivalence approach using the following standards: the ratio of geometric LSmeans with corresponding 90% confidence interval calculated from the exponential of the difference between the Test and the Reference for the ln-transformed parameters Cmax and AUC0-T should all be within the 80.00 to 125.00% bioequivalence range.

The safety population will include all subjects who received at least one dose of one of the IPs. Safety assessments will include clinical laboratory tests, and adverse event (AE) monitoring. Additional safety measurements may be performed at the discretion of the investigator for reasons related to subject safety. The physician in charge will be present at the clinical site for at least the first 4 hours following each drug administration and will remain available at all times throughout the study.

Total study duration: up to 35 days (including screening).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Healthy male or female adult volunteer
4. A female volunteer meeting one of the following criteria:

   1. Participant is of childbearing potential and agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first study drug administration through to at least 30 days after the last dose of the study drug. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse
      * Systemic contraceptives (combined birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
      * Intrauterine device (IUD) (with or without hormones)
      * Male condom with spermicide or male condom with a vaginal spermicide (gel, foam, or suppository)
      * Male partner vasectomized at least 6 months prior to the first study drug administration

      Or
   2. Participant whose partner has had a vasectomy less than 6 months prior to dosing, and agrees to use an additional acceptable method of contraception from the first study drug administration through to at least 30 days after the last dose of the study drug

      Or
   3. Participant is of non-childbearing potential, defined as surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is in a postmenopausal state (i.e. at least 1 year without menses without an alternative medical condition prior to the first study drug administration)
5. Volunteer aged at least 18 years
6. Volunteer with a body mass index (BMI) within 18.5 kg/m2 to 30.0 kg/m2, inclusively
7. Non- or ex-smoker; an ex-smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration
8. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without clinical significance, as determined by an investigator
9. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an investigator

Exclusion Criteria:

1. Females who are lactating at screening
2. Females who are pregnant according to the pregnancy test at screening or prior to the first study drug administration
3. History of significant hypersensitivity to febuxostat or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
4. Presence of significant gastrointestinal, liver or kidney disease, or any other condition known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects
5. History of significant gastrointestinal, liver or kidney disease that may affect drug bioavailability
6. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
7. Presence of clinically significant ECG abnormalities at the screening visit, as defined by medical judgment
8. History of rare hereditary problems of galactose and/or lactose intolerance, lactase deficiency or glucose-galactose malabsorption
9. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
10. Any clinically significant illness in the 28 days prior to the first study drug administration
11. Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) in the 28 days prior to the first study drug administration, that in the opinion of an investigator would put into question the status of the volunteer as healthy
12. Any history of tuberculosis
13. Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration
14. Positive screening results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG (B) (hepatitis B)) or Hepatitis C Virus (HCV (C)) tests
15. Volunteers who have already been included in a previous group for this clinical study
16. Volunteers who took febuxostat in the 28 days prior to the first study drug administration
17. Volunteers who took an Investigational Product (IP) in the 28 days prior to the first study drug administration
18. Volunteers who donated 50 mL or more of blood in the 28 days prior to the first study drug administration
19. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Cmax of febuxostat in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.25, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 18.00, 24.00, 36.00 hours after each drug administration
  Maximum observed concentration in plasma
AUC0-T of febuxostat in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.25, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 18.00, 24.00, 36.00 hours after each drug administration
  Cumulative area under the concentration time curve calculated from 0 to time of last observed quantifiable concentration (TLQC) using the linear trapezoidal method

SECONDARY OUTCOMES:
Tmax of febuxostat in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.25, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 18.00, 24.00, 36.00 hours after each drug administration
  Time of maximum observed concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value
TLQC of febuxostat in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.25, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 18.00, 24.00, 36.00 hours after each drug administration
  Time of last observed quantifiable concentration
AUC0-∞ of febuxostat in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.25, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 18.00, 24.00, 36.00 hours after each drug administration
  Area under the concentration time curve extrapolated to infinity, calculated as AUC0-T + ĈLQC (the predicted concentration at time TLQC) / λZ (apparent elimination rate constant)
Residual area of febuxostat in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.25, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 18.00, 24.00, 36.00 hours after each drug administration
  Extrapolated area (i.e. percentage of AUC0-∞ due to extrapolation from TLQC to infinity)
Time point where the log-linear elimination phase begins (TLIN) of febuxostat in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.25, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 18.00, 24.00, 36.00 hours after each drug administration
  Time point where the log-linear elimination phase begins
λZ of febuxostat in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.25, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 18.00, 24.00, 36.00 hours after each drug administration
  Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration versus time curve
Terminal elimination half-life (Thalf) of febuxostat in plasma after administration of the test and the reference products | Time points 0.00 (prior to each drug administration) and 0.25, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 2.00, 2.50, 3.00, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 15.00, 18.00, 24.00, 36.00 hours after each drug administration
  Terminal elimination half-life, calculated as ln(2)/λZ
Number of treatment-emergent adverse events for the test and the reference products | Up to 9 days (after the first drug administration until the completion of clinical part of the study)]
  The safety population will include all subjects who received at least one dose of the test or the reference product. Any significant changes will be recorded as treatment-emergent adverse events only if they are judged clinically significant by the qualified investigator or delegate.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Altasciences Company Inc.
Locations (1):
- Altasciences Company Inc., Montreal, Quebec, Canada